CLINICAL TRIAL: NCT06622330
Title: The Effect of Position Change on Pain and Cerebral Oxygen Saturation After Endotracheal Aspiration
Brief Title: The Effect of Position Change on Pain and Cerebral Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Ph.D., Asst. Prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-15916306-604.01.01-209306724
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Children
Keywords: Pediatrics; position; pain; oxygen saturation
MeSH Terms: conditions — Pain | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group given position (Experimental): Children in the experimental group were given 30 minutes of wrapping and 30 minutes of fetal position after aspiration.
  Interventions: Other: Positioning
- Control group (No Intervention): No intervention was made to the control group.

INTERVENTIONS:
Other: Positioning — Children in the experimental group were given 30 minutes of wrapping and 30 minutes of fetal position after aspiration.
  Arms: Group given position

SUMMARY:
This study is a randomized controlled experimental study to investigate the effect of position change on pain and cerebral oxygen saturation after endotracheal aspiration in pediatric patients.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental study to investigate the effect of position change on pain and cerebral oxygen saturation after endotracheal aspiration in pediatric patients. The study sample consisted of 70 pediatric patients (35 in the control group and 35 in the intervention group) who met the inclusion criteria and whose parents gave informed consent. The research data were collected using the "Child Identification Form" and the "Behavioral Pain Scale". SPSS 24 program was used to analyze the data obtained in the study. Children in the experimental group were given 30 minutes of wrapping and 30 minutes of fetal position after aspiration. Children in the control group did not receive any treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients whose consent form is signed by their legal guardian
* Intubated pediatric patients receiving mechanical ventilation support
* Non-sedatized pediatric patients
* Pediatric patients who have received only paracetamol and whose duration of action has exceeded 4-6 hours

Exclusion Criteria:

* Unconscious pediatric patients
* Pediatric patients receiving pharmacologic drugs other than paracetamol
* Unstable pediatric patients
* Pediatric patients with painful procedures during the procedure

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Behavioral Pain Scale | Measured before aspiration, 1 and 2 hours after aspiration. Each measurement lasted 10 minutes.
  Determines the pain level of children. In this scale, there are three items including facial expression, upper extremities and ventilator compliance and four variables including behavioral responses to pain in each item. These are; facial expression (relaxed, partially relaxed, fully tense, grimace), upper extremities (no movement, partially flexed, fully flexed), fingers (flexed, continuously retracted), compliance with ventilation (tolerates ventilation, coughs, but often tolerates ventilation, fights with ventilator, cannot control ventilation). Each question is given a score between 1-4. The lowest score is 3 and the highest score is 12. The higher the score, the more severe the pain.
Cerebral oxygen saturation | Measured before aspiration, 1 and 2 hours after aspiration. Each measurement lasted 10 minutes.
  It was measured to determine the cerebral oxygen saturation of children.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kökcü Doğan, Study Director — 444 85 44; Aysel Kökcü Doğan, Study Director — Istanbul Medipol UniversityInstitute of Health Sciences
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)